CLINICAL TRIAL: NCT01891279
Title: The Use of Elemental Formula in Neonates Post Small Bowel Resection: Improved Success to Wean From Total Parenteral Nutrition?
Brief Title: Elemental Formula in Neonates Post Small Bowel Resection: Improved Weaning From Total Parenteral Nutrition?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Amir Mustafa Khan, Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HSC-MS-09-0260
Record Dates: First submitted 2012-05-01; First posted 2013-07-03 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: short bowel syndrome; Elemental formula; partially hydrolyzed formula; Enteral feeding; TPN dependency; Intestinal adaptation; TPN cholestasis
MeSH Terms: conditions — Short Bowel Syndrome | interventions — pregestimil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- elemental formula, Elecare® (Experimental): Babies will receive elemental formula, Elecare®, if breast milk is not available.
  Interventions: Other: elemental formula Elecare®
- part hydrolyzed formula, Pregestimil® (Experimental): Babies will receive partially hydrolyzed formula, Pregestimil®, if breast milk is not available.
  Interventions: Other: partially hydrolyzed formula

INTERVENTIONS:
Other: elemental formula Elecare® — Babies will be randomized to received either elemental formula (Elecare®) or partially hydrolyzed formula (Pregestimil®) if breast milk is not available.
  Other Names: Elecare®
  Arms: elemental formula, Elecare®
Other: partially hydrolyzed formula — Babies will be randomized to received either partially hydrolyzed formula (Pregestimil®) or elemental formula (Elecare®)if breast milk is not available.
  Other Names: Pregestimil®
  Arms: part hydrolyzed formula, Pregestimil®

SUMMARY:
In neonates with recent small bowel resection or congenital bowel anomalies (gastroschisis or omphalocele), does an elemental formula as compared to a partially hydrolyzed formula allowed the infant to wean off Total Parenteral Nutrition (TPN) earlier?

DETAILED DESCRIPTION:
Neonates with short bowel syndrome (SBS) due to recent small bowel resection or congenital bowel anomalies (gastroschisis or omphalocele) can have inability to adequately digest and absorb enteral feedings resulting in prolonged Parenteral Nutrition (PN) dependence for nutrition and growth. Prolonged PN dependence can result in Parenteral Nutrition Associated Liver Disease (PNALD) and intestinal failure requiring small bowel or small bowel/liver transplantation for survival.

After bowel resection, the bowel has an ability to compensate for significant loss by going through a process called intestinal adaptation. Enteral feeding is the key factor for initiating and maintaining the adaptation of the intestine.

Whole protein formulas or partially hydrolyzed formulas provide either the full protein or dipeptides/tripeptides respectively, and are thought to confer the best benefit in inducing intestinal adaptation and increasing paracrine stimulation. However, in small studies of adults and children with SBS,an amino acid based (elemental) formula demonstrated improved feeding tolerance and ability to wean off TPN. In a small study, babies fed breast milk or elemental formula appeared to have shorter duration of TPN.

This is a randomized, blinded clinical trial to determine if elemental formula, Elecare® (vs. partially hydrolyzed formula, Pregestimil®) is better tolerated and allows a higher proportion of neonates with small bowel resection or congenital bowel anomalies to successfully wean off TPN.

ELIGIBILITY:
Inclusion Criteria:

* Term or pre-term neonates with either surgical resection of the small bowel or congenital bowel anomalies (gastroschisis, omphalocele) unable to tolerate 90kcal/kg/day of enteral feedings by 1 month of age

Exclusion Criteria:

* Term or preterm neonates with NEC totalis,
* Inborn Errors of Metabolism, or
* Known or suspected congenital syndromes

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2011-09-26 (Actual); Primary Completion 2013-08-13 (Actual); Study Completion 2013-09-17 (Actual)

PRIMARY OUTCOMES:
tolerance of TPN use | 6 weeks and 8 weeks after initiation of feeding
  At 6 wks post intervention, if they are tolerating < 40 enteral Kcal/k/day, this will be considered a failure to establish adaptation with the formula; if they are tolerating 41-90 enteral Kcal/k/day, this formula will be continued for 2 weeks longer;if they are tolerating >90 enteral Kcal/k/day, this will be considered a weaning success.
  At 8 wks post intervention, if they are tolerating <90 enteral Kcal/k/day, this will be considered a failure to establish adaptation; At 8 wks post intervention, if they are tolerating >90 enteral Kcal/k/day, this will be considered a weaning success.

SECONDARY OUTCOMES:
Length of hospital stay | from birth (admission) to discharge (up to 1 year of age)
  number of hospital days from birth to hospital discharge, up to 1 year of age
Direct bilirubin levels | From birth (admission) to discharge (up to 1 year of age)
  The highest and lowest direct bilirubin levels during hospitalization and direct bilirubin level at hospital discharge
Blood stream infections | From birth (admission) to discharge (up to 1 year of age)
  Assessment for signs of infection (e.g. CBC, CRP, blood cultures, UA, stool studies, C. diff) is routine.

CONTACTS AND LOCATIONS:
Overall Officials: Amir M Khan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Vanderhoof JA. Short bowel syndrome in children and small intestinal transplantation. Pediatr Clin North Am. 1996 Apr;43(2):533-50. doi: 10.1016/s0031-3955(05)70419-3. PMID 8614614
- [Background] Vanderhoof JA. Short bowel syndrome. Clin Perinatol. 1996 Jun;23(2):377-86. PMID 8780910
- [Background] Bines JE, Taylor RG, Justice F, Paris MC, Sourial M, Nagy E, Emselle S, Catto-Smith AG, Fuller PJ. Influence of diet complexity on intestinal adaptation following massive small bowel resection in a preclinical model. J Gastroenterol Hepatol. 2002 Nov;17(11):1170-9. doi: 10.1046/j.1440-1746.2002.02872.x. PMID 12453276
- [Background] Bines J, Francis D, Hill D. Reducing parenteral requirement in children with short bowel syndrome: impact of an amino acid-based complete infant formula. J Pediatr Gastroenterol Nutr. 1998 Feb;26(2):123-8. doi: 10.1097/00005176-199802000-00001. PMID 9481624
- [Background] Lai HS, Chen WJ, Chen KM, Lee YN. Effects of monomeric and polymeric diets on small intestine following massive resection. Taiwan Yi Xue Hui Za Zhi. 1989 Oct;88(10):982-8. PMID 2634733
- [Background] Cosnes J, Evard D, Beaugerie L, Gendre JP, Le Quintrec Y. Improvement in protein absorption with a small-peptide-based diet in patients with high jejunostomy. Nutrition. 1992 Nov-Dec;8(6):406-11. PMID 1486247
- [Background] Andorsky DJ, Lund DP, Lillehei CW, Jaksic T, Dicanzio J, Richardson DS, Collier SB, Lo C, Duggan C. Nutritional and other postoperative management of neonates with short bowel syndrome correlates with clinical outcomes. J Pediatr. 2001 Jul;139(1):27-33. doi: 10.1067/mpd.2001.114481. PMID 11445790
- [Background] Rhoads JM, Plunkett E, Galanko J, Lichtman S, Taylor L, Maynor A, Weiner T, Freeman K, Guarisco JL, Wu GY. Serum citrulline levels correlate with enteral tolerance and bowel length in infants with short bowel syndrome. J Pediatr. 2005 Apr;146(4):542-7. doi: 10.1016/j.jpeds.2004.12.027. PMID 15812462
- [Background] Jianfeng G, Weiming Z, Ning L, Fangnan L, Li T, Nan L, Jieshou L. Serum citrulline is a simple quantitative marker for small intestinal enterocytes mass and absorption function in short bowel patients. J Surg Res. 2005 Aug;127(2):177-82. doi: 10.1016/j.jss.2005.04.004. PMID 15921697
- [Background] Crenn P, Vahedi K, Lavergne-Slove A, Cynober L, Matuchansky C, Messing B. Plasma citrulline: A marker of enterocyte mass in villous atrophy-associated small bowel disease. Gastroenterology. 2003 May;124(5):1210-9. doi: 10.1016/s0016-5085(03)00170-7. PMID 12730862
- [Background] Crenn P, Coudray-Lucas C, Thuillier F, Cynober L, Messing B. Postabsorptive plasma citrulline concentration is a marker of absorptive enterocyte mass and intestinal failure in humans. Gastroenterology. 2000 Dec;119(6):1496-505. doi: 10.1053/gast.2000.20227. PMID 11113071